CLINICAL TRIAL: NCT02298270
Title: Resiliency Training for Patients With Neurofibromatosis Via Videoconferencing With Skype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Children's Tumor Foundation (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Dr., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013P002605a
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Neurofibromatosis; Neurofibromatosis I; Neurofibromatosis 2; Schwannomatosis
Keywords: Neurofibromatosis; NF I; NF 2; Schwannomatosis; Stress Management; Resiliency; Skype
MeSH Terms: conditions — Neurofibromatoses; Neurofibromatosis 1; Neurofibromatosis 2; Schwannomatosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation Response Resiliency Program (Experimental): Participants will receive an 8-week behavioral intervention which teaches stress management and psychological resiliency-enhancing skills.
  Interventions: Behavioral: The Relaxation Response Resiliency Program (3RP) via Skype
- Health Education (Placebo Comparator): Participants will receive and 8-week general stress and health education program, with none of the active relaxation and resiliency-based components being tested in the experimental condition.
  Interventions: Behavioral: The Relaxation Response Resiliency Program (3RP) via Skype

INTERVENTIONS:
Behavioral: The Relaxation Response Resiliency Program (3RP) via Skype — 8-week group intervention, delivered via Skype, teaching relaxation and psychological resiliency enhancing skills. Topics include the relaxation response, meditation, and yoga.

SUMMARY:
This study tests the efficacy of an 8-week, Skype-based, group resiliency training intervention (The Relaxation Response Resiliency Program) for improving psychological stress in patients with Neurofibromatosis. A control group will receive a general health education curriculum. The investigators hypothesize that patients will improve on measures of psychological stress as a result of the resiliency program.

A substudy (Unique Protocol ID: 2013P002605b) has been approved to test this study on a sub-population: patients with NF2 who are hard of hearing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Can read and speak English at or above the 6th grade level
3. Diagnosis of neurofibromatosis type 1, neurofibromatosis type 2, or schwannomatosis

Exclusion Criteria:

1. Severe active or untreated major mental illness that would interfere with study participation, to be determined at the discretion of the study investigator (e.g. untreated psychosis or suicidality)
2. Recent (within past 3 months) change in antidepressant medication
3. Use of formal relaxation training (including past participation in a mind-body program), currently or in the past 6 months.
4. Unable or unwilling to sign the informed consent documents
5. Unable or unwilling to complete psychological assessments online via the REDCap system.
6. Unable or unwilling to participate in an intervention delivered via videoconferencing with Skype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Life (SWL) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Satisfaction with Life (SWL) scale is a reliable and valid 5-item self-report measure of global life satisfaction. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.
Quality of Life (WHOQOL-BREF) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The WHOQOL-BREF comprises of 26 items which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PSS is a widely used psychological instrument for the measurement of the perception of stress. This 10-itam scale is designed to measure the degree to which situations in one's life are appraised, or considered stressful. The scores range from 0-40, with a higher score indicating higher perceived stress. Items were designed to detect how unpredictable, uncontrollable and overloaded respondents find their lives.
The Pain Catastrophizing Scale (PCS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Pain Catastrophizing Scale (PCS) is widely used to assess cognitive and affective responses to pain and to evaluate pain management program outcomes.
Pain Numerical Rating Scale (Pain NRS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Pain NRS is a scale for patient self-reporting measurements of pain. The measure was depicted by REINS as a standard measure to use in Neurofibromatosis clinical trials.
Patient Health Quesionnaire (PHQ) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PHQ measures symptoms of depression and functional impairment.
Brief Pain Inventory (BPI) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Brief Pain Inventory (BPI) allows patients to rate the severity of their pain (BPI-S) and the degree to which their pain interferes with common dimensions of feeling and function (BPI-I).
Cognitive and Affective Mindfulness Scale (CAMS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The CAMS measures the degree to which individuals experience their thoughts and feelings.
Posttraumatic Growth Inventory (PGI) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PGI is an instrument for assessing positive outcomes reported by persons who have experienced traumatic events.
Interpersonal Reactivity Index (IRI) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The IRI assesses the cognitive and affective dimensions of empathy.
Distress Analogue Scales | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32). Also administered at mid-interevention, before each group session.
  The Distress Analogue Scales measure participants' levels of stress, coping, distress, and discomfort.
Epworth Sleepiness Scale (ESS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Epworth Sleepiness Scale (ESS) has been widely used to assess a person's average level of daytime sleepiness in daily life.
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOCS-A is a 13-item measure assessing participants' current self-perceived status on several skills such as: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.
Life Orientation Test (LOT) Optimism Scale | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The LOT Optimism Scale measures individual differences in generalized optimism versus pessimism.
The Gratitude Questionnaire (GQ-6) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The GQ-6 revised is a 6-item measure that assesses individual differences in the proneness to experience gratitude in daily life. Scores range from 6-42, with a higher score indicating a greater sense of gratitude.
Functional Assessment of Chronic Illness Therapy- Fatigue Scale (FACIT-Fatigue) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The FACIT-Fatigue measures participants' tiredness, weakness, and difficulty conducting usual activities due to fatigue.
Functional Assessment of Chronic Illness Therapy- Spirituality Scale (FACIT-Sp) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The FACIT-Sp measures participants' spiritual well-being (sense of meaning in life and the sense of strength in one's faith) over the past 7 days.
Medical Outcomes Study (MOS) Social Support Survey | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOS Social Support Survey measures various dimensions of social support.
The 14-Item Resiliency Scale (RS-14) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The RS-14 measures stress coping ability in the face of adversity.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States